CLINICAL TRIAL: NCT04231838
Title: A Randomised Controlled International Multicentre Study Evaluating Changes in Metabolic Syndrome in Smokers With Type 2 Diabetes Mellitus After Switching From Tobacco Cigarettes to Combustion-Free Nicotine Delivery Systems: DIASMOKE Study
Brief Title: Metabolic Syndrome in Diabetic Smokers Using Cigarettes & Combustion-Free Nicotine Delivery Systems
Acronym: DIASMOKE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eclat Srl. (Other)
Collaborators: University of Catania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: COE1-05-DIASMOKE 2.0
Record Dates: First submitted 2019-12-11; First posted 2020-01-18 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Cardiovascular Risk Factor; Diabetes Mellitus, Type 2
Keywords: e-cigarettes; Combustion-Free Nicotine Delivery Systems; Diabetes Mellitus, Type 2; Cardiovascular Risk Factor; Tobacco Cigarettes; DIASMOKE 2.0; Metabolic syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Vaping; Metabolic Syndrome | interventions — Tobacco Products

STUDY DESIGN:
Intervention Model Description: Study Arms and Randomization Plan Participants who were eligible and consent to take part will be randomized to either continuing smoking their own cigarette brand (Arm A) or switching to using C-F NDS (Arm B).
  The randomization sequence will be computer generated, with an allocation ratio of 1:2 (Arm A: Arm B) to compensate for an estimated 50% success rate (defined as combined smoking abstinence rate + >80% smoking reduction rate) in the long term (more details in the section about Sample Size Calculation). The randomization scheme will be provided to clinical sites via a web-based application set up by the CRO. The staff randomizing the participant will access the web-based application when the participant is with them, entering their participant identification number, date of birth and initials into the program. The allocation will be immediately provided by the program/software.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Arm (Arm A) (Active Comparator): Participant continues smoking their own cigarette brand.
  Interventions: Other: TOBACCO CIGARETTES
- Intervention Arm (Arm B) (Active Comparator): Participant switches to using C-F NDS
  Interventions: Other: COMBUSTION-FREE NICOTINE DELIVERY SYSTEMS (C-F NDS)

INTERVENTIONS:
Other: TOBACCO CIGARETTES — Participants in Arm A will continue smoking their own cigarette brand as usual.
  Arms: Standard Arm (Arm A)
Other: COMBUSTION-FREE NICOTINE DELIVERY SYSTEMS (C-F NDS) — Participants in Arm B will trial and familiarize with their allocated products to select the C-F NDS of their preference. They will be trained and counselled on the chosen C-F NDS; participants will also have the option to try and choose among a selection of either 3 e-liquids or 3 tobacco sticks (depending on the C-F NDS they have chosen). Participants wishing to use a heated tobacco device (HTD) will receive one kit and a full 1 week supply of tobacco sticks of their choice (they will receive a number of tobacco sticks/day corresponding to the number of cigarettes smoked at baseline); those wishing to use a vaping product will receive one vaping kit and a full 1 week supply of e-liquids of their choice (they will receive 4 x 10 ml refill containers).
  Arms: Intervention Arm (Arm B)

SUMMARY:
Very little is known about the impact of combustion-free nicotine delivery systems (C-F NDS) on cardiovascular risk factors in T2DM patients who smoke. Data from clinical studies to identify any potential reduction in individuals' risk, relative to the risk of continued smoking, are needed.

This study aims to test the hypothesis that avoiding exposure to cigarette smoke toxicants may translate to measurable improvement in cardiovascular risk factors and functional parameters when T2DM patients who smoke switch to using C-F NDS compared with T2DM patients who continue to smoke conventional tobacco products.

The investigators propose a prospective 2-year multicenter randomized controlled trial (RCT) to evaluate changes in cardiovascular risk factors and functional parameters in diabetic smokers using C-F NDS and compared to those continuing cigarette smoking.

DETAILED DESCRIPTION:
This is a multicenter, controlled study utilizing a randomized switching design for cigarette smoking and C-F NDS use. The study will take place in one site in each of five countries. Three countries have so far agreed to participate: UK, Italy, Poland. An amendment will be submitted to the REC once the final two countries are signed up.

A volunteer population of adult smokers with T2DM will be recruited. Smokers will be randomized (1:2 ratio) to either continue to smoke their own cigarette brand (Study Arm A) or use C-F NDS (Study Arm B). The intended minimum number of participants in each arm by the end of the study is 147.

Before randomization, all smokers will be reminded of the risks associated with smoking and will be offered a free smoking cessation program according to standard local guidelines and depending on the local availability of antismoking services. Those who decline the invitation will be eligible for recruitment into the RCT.

Smokers are free to voluntarily quit smoking/C-F NDS and/or withdraw from the study at any time.

Duration:

This will be a prospective 2-year study conducted in the ambulatory setting. Participants will attend a total of 5 clinic visits at Screening, Day 1 (Visit 1), Day 90 (+/-5 days) (Visit 2), Day 180 (+/-7 days) (Visit 3), Day 360 (+/-7 days) (Visit 4), and Day 720 (+/-7 days) (Visit 5).

Participants will undergo screening within 28 days prior to Day 1. Eligible participants will be enrolled and randomized on Day 1.

Study Arms and Randomization Plan Participants who were eligible and consent to take part will be randomized to either continuing smoking their own cigarette brand (Arm A) or switching to using C-F NDS (Arm B).

The randomization sequence will be computer generated, with an allocation ratio of 1:2 (Arm A: Arm B) to compensate for an estimated 50% success rate (defined as combined smoking abstinence rate + >80% smoking reduction rate) in the long term (more details in the section about Sample Size Calculation). The randomization scheme will be provided to clinical sites via a web-based application set up by the CRO. The staff randomizing the participant will access the web-based application when the participant is with them, entering their participant identification number, date of birth and initials into the program. The allocation will be immediately provided by the program/software.

Product Use Smokers will continue to smoke their usual brand of cigarette until randomization on Day 1. After randomization, participants in Arms A and B will be asked to use only their assigned products ad libitum for the whole duration of the study (for more info/details - see below).

Participants in Arm A will continue smoking their own cigarette brand as usual. Participants in Arm B will trial and familiarize with their allocated products to select the C-F NDS of their preference. They will be trained and counseled on the chosen C-F NDS; participants will also have the option to try and choose among a selection of either 3 e-liquids or 3 tobacco sticks (depending on the C-F NDS they have chosen). Participants wishing to use a heated tobacco device will receive one kit and a full 1 week supply of tobacco sticks of their choice (they will receive a number of tobacco sticks/day corresponding to the number of cigarettes smoked at baseline); those wishing to use a vaping product will receive one vaping kit and a full 1 week supply of e-liquids of their choice (they will receive 4, 10 ml refill containers). Free products will be supplied at each subsequent visit throughout the whole duration of the study

Product Monitoring and Compliance A prospective evaluation of cigarette consumption will be carried out throughout the study (see below). Cigarette use will be self-reported and recorded in the eCRF/ automated eDiary-SMS system (+ APP tracker).

Participants in Arm B will be instructed on the importance of using exclusively their C-F NDS and to abstain from smoking. Participants will be asked to report any non-compliance via the automated eDiary-SMS system (+ APP tracker), and will be informed that compliance assessments will be conducted throughout the study. Non-compliance will be documented.

Justification for Study Design

Participants in this study will be a minimum of 23 years of age. This is based on:

* The legal age to obtain tobacco products is 18 years
* Participants will be required to have a smoking history of at least 5 years To investigate the effects of abstaining from smoking by switching in smokers with T2DM, a population of patients who are intending to make the switch to N-C NDS will be recruited. By the end of the study, it is estimated that a high proportion (approx. 50%) of patients randomized in the Arm B of the study will not be able to achieve success (defined as either complete smoking abstinence or as at least 80% smoking reduction). To account for this, the C-F NDS population will be oversampled and a 1:2 randomization ratio scheme (i.e. for every patient randomized in the continue-to-smoke population, two will be randomized in the C-F NDS population) will be adopted.

Treatment blinding This is an unblinded study. It will not be possible to blind participants to the intervention they will be receiving. It will not be possible to blind trial staff when providing the interventions and collecting data.

Unblinded data will be seen and analysed by the Trial Statistician for the purposes of the Data Monitoring and Ethics Committee (DMEC) meetings. All other trial staff who has access to outcome data will remain blinded until prespecified data analyses will be completed. Prespecified data analyses will be conducted blind to treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

Participants will be required to satisfy all of the following criteria at the screening visit, unless otherwise stated:

• Participants will be: 1.1. over 23 years of age

• T2DM Patients will have: 2.1. body mass index (BMI) between 17.6 and 34.5 kg/m2, inclusive 2.2. body weight exceeding 50 kg (males) or 40 kg (females) 2.3 6.0<HbA1C<12 3.2. completion of proforma (CRF) 3.3. lab assessment as outlined in the CRF

* Participants will be willing to refrain from eating/drinking prior to screening and Check-in at each study visit.
* Participants will be regular smokers of at least 10 cigarettes/day (max 30 cigarette/day)
* Participants will have smoked for at least five consecutive years prior to screening.
* Participants must have a saliva cotinine level > 10 ng/mL or an exhaled breath CO (eCO) level > 7 ppm at screening.
* Participants in Arm A who continue to smoke will be willing to use their own brand/type cigarettes.
* Participants in Arms B will be willing to use the study products (THP product or e-cigarette) provided to them during the study.

Exclusion Criteria:

Participants will be excluded at the screening visit based on the following criteria:

* Female participants who are pregnant or breastfeeding. This will be confirmed at screening and at visit 1. Any female subject who becomes pregnant during this study will be withdrawn.
* Participants with a history of recent acute decompensation of their disease requiring treatment within 4 weeks prior to visit 1.
* Participants who have a significant history of alcoholism or drug/chemical abuse within 24 months prior to screening, as determined by the investigator.
* Participants who are still participating in another clinical study (e.g. attending follow-up visits) or who have participated in a clinical study involving administration of an investigational drug (new chemical entity) in the past 3 months prior to first product use.
* Participants who have, or who have a history of, any clinically-significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, haematological or other major disorder that, in the opinion of the investigator or their appropriately qualified designee, would jeopardise the safety of the subject or impact on the validity of the study results.
* Participants who regularly use any nicotine (e.g. e-cigarettes, NRT) or tobacco product (e.g. HTPs, oral smokeless) other than their own cigarettes within 14 days of screening.

At screening and prior to enrolment, all patients will be offered a locally available free smoking cessation program as per local guidelines. Those who express the intention of booking for the cessation program together with those who, at screening, are planning to quit smoking in the next 6 months, will not be recruited in the study. Patients taking part in the study will be informed that they are free to quit smoking and withdraw from the study at any time. Any subject who decides to quit smoking will be directed to local stop smoking services.

Withdrawal Criteria:

Patients may be withdrawn from the study prematurely for the following reasons:

1. subject experiences a severe adverse event (SAE). The appropriate SAE electronic Case Report Form (eCRF) page must be completed.
2. If any deviations occur during the conduct of the study, which cannot be corrected. All protocol deviations will be fully documented and considered for their effect on study objectives. Deviations that could lead to subject discontinuation from the study include:

   * deviations which could affect subject's safety (e.g. illness requiring treatment[s]) which in the clinical judgement of the investigator might invalidate the study by interfering with the allocated test product or the willingness of the subject to comply with the study activities.
   * deviations involving the use of any nicotine/tobacco products other than the intended conventional cigarettes (in Arm A) or (in Arm B).
3. If the subject is uncooperative, including non-attendance. In these cases, efforts should have been made by the investigator to ascertain the reason and to ensure the subject's attendance as soon as possible.
4. Subject's personal request: the subject could decide, at any moment of the study, to stop his/her participation.
5. Female participant becoming pregnant.

Min Age: 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2025-09-16 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Metabolic Syndrome Prevalence | Changes in the prevalence of Metabolic Syndrome from baseline will be assessed at 3 months, 6 months, 1 year, and 2 years
  Percentage (%) change in Metabolic Syndrome Prevalence

SECONDARY OUTCOMES:
Change in Plasma Glucose | Change in plasma glucose from baseline will be assessed at 3 months, 6 months, 1 year, and 2 years
  Change in plasma glucose (mmol/L) will be measured from baseline at different study time-points
Change in Blood Pressure | Change in blood pressure from baseline will be assessed at 3 months, 6 months, 1 year, and 2 years
  Change in blood pressure (mmHg) will be measure from baseline at different study time-points
Change in Triglycerides | Change in triglycerides from baseline will be assessed at 3 months, 6 months, 1 year, and 2 years
  Change in triglycerides (mmol/L) will be measured from baseline at different study time-points
Change in High-Density Lipoprotein (HDL) | Change in HDL from baseline will be assessed at 3 months, 6 months, 1 year, and 2 years
  Change in HDL (mmol/L) will be measured from baseline at different study time-points
Change in Waist Circumference | Change in waist circumference from baseline will be assessed at 3 months, 6 months, 1 year, and 2 years
  Change in waist circumference (cm) will be measured from baseline at different study time-points

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Sharma, PhD, Principal Investigator — Ashford and St Peter's Hospitals NHS Foundation Trust
Locations (1):
- Ashford and St Peters NHS Foundation Trust, Chertsey, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fowler MJ. Microvascular and Macrovascular Complications of Diabetes. Clinical Diabetes. 2011;29:116-22.
- [Background] Pan A, Wang Y, Talaei M, Hu FB, Wu T. Relation of active, passive, and quitting smoking with incident type 2 diabetes: a systematic review and meta-analysis. Lancet Diabetes Endocrinol. 2015 Dec;3(12):958-67. doi: 10.1016/S2213-8587(15)00316-2. Epub 2015 Sep 18. PMID 26388413
- [Background] Wei M, Gaskill SP, Haffner SM, Stern MP. Effects of diabetes and level of glycemia on all-cause and cardiovascular mortality. The San Antonio Heart Study. Diabetes Care. 1998 Jul;21(7):1167-72. doi: 10.2337/diacare.21.7.1167. PMID 9653614
- [Background] Al-Delaimy WK, Manson JE, Solomon CG, Kawachi I, Stampfer MJ, Willett WC, Hu FB. Smoking and risk of coronary heart disease among women with type 2 diabetes mellitus. Arch Intern Med. 2002 Feb 11;162(3):273-9. doi: 10.1001/archinte.162.3.273. PMID 11822919
- [Background] Chuahirun T, Simoni J, Hudson C, Seipel T, Khanna A, Harrist RB, Wesson DE. Cigarette smoking exacerbates and its cessation ameliorates renal injury in type 2 diabetes. Am J Med Sci. 2004 Feb;327(2):57-67. doi: 10.1097/00000441-200402000-00001. PMID 14770020
- [Background] Qin R, Chen T, Lou Q, Yu D. Excess risk of mortality and cardiovascular events associated with smoking among patients with diabetes: meta-analysis of observational prospective studies. Int J Cardiol. 2013 Jul 31;167(2):342-50. doi: 10.1016/j.ijcard.2011.12.100. Epub 2012 Jan 16. PMID 22251416
- [Background] Pan A, Wang Y, Talaei M, Hu FB. Relation of Smoking With Total Mortality and Cardiovascular Events Among Patients With Diabetes Mellitus: A Meta-Analysis and Systematic Review. Circulation. 2015 Nov 10;132(19):1795-804. doi: 10.1161/CIRCULATIONAHA.115.017926. Epub 2015 Aug 26. PMID 26311724
- [Background] Cacciola RR, Guarino F, Polosa R. Relevance of endothelial-haemostatic dysfunction in cigarette smoking. Curr Med Chem. 2007;14(17):1887-92. doi: 10.2174/092986707781058832. PMID 17627524
- [Background] Stanton CA, Keith DR, Gaalema DE, Bunn JY, Doogan NJ, Redner R, Kurti AN, Roberts ME, Higgins ST. Trends in tobacco use among US adults with chronic health conditions: National Survey on Drug Use and Health 2005-2013. Prev Med. 2016 Nov;92:160-168. doi: 10.1016/j.ypmed.2016.04.008. Epub 2016 Apr 15. PMID 27090919
- [Background] Ford ES, Mokdad AH, Gregg EW. Trends in cigarette smoking among US adults with diabetes: findings from the Behavioral Risk Factor Surveillance System. Prev Med. 2004 Dec;39(6):1238-42. doi: 10.1016/j.ypmed.2004.04.039. PMID 15539062
- [Background] Caponnetto P, Russo C, Polosa R. Smoking cessation: present status and future perspectives. Curr Opin Pharmacol. 2012 Jun;12(3):229-37. doi: 10.1016/j.coph.2012.02.005. Epub 2012 Mar 5. PMID 22398322
- [Background] Polosa R, Benowitz NL. Treatment of nicotine addiction: present therapeutic options and pipeline developments. Trends Pharmacol Sci. 2011 May;32(5):281-9. doi: 10.1016/j.tips.2010.12.008. Epub 2011 Jan 20. PMID 21256603
- [Background] Nagrebetsky A, Brettell R, Roberts N, Farmer A. Smoking cessation in adults with diabetes: a systematic review and meta-analysis of data from randomised controlled trials. BMJ Open. 2014 Mar 6;4(3):e004107. doi: 10.1136/bmjopen-2013-004107. PMID 24604481
- [Background] Polosa R, Rodu B, Caponnetto P, Maglia M, Raciti C. A fresh look at tobacco harm reduction: the case for the electronic cigarette. Harm Reduct J. 2013 Oct 4;10:19. doi: 10.1186/1477-7517-10-19. PMID 24090432
- [Background] Farsalinos KE, Polosa R. Safety evaluation and risk assessment of electronic cigarettes as tobacco cigarette substitutes: a systematic review. Ther Adv Drug Saf. 2014 Apr;5(2):67-86. doi: 10.1177/2042098614524430. PMID 25083263
- [Background] Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults. Executive Summary of The Third Report of The National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, And Treatment of High Blood Cholesterol In Adults (Adult Treatment Panel III). JAMA. 2001 May 16;285(19):2486-97. doi: 10.1001/jama.285.19.2486. No abstract available. PMID 11368702
- [Background] Metascreen Writing Committee; Bonadonna R, Cucinotta D, Fedele D, Riccardi G, Tiengo A. The metabolic syndrome is a risk indicator of microvascular and macrovascular complications in diabetes: results from Metascreen, a multicenter diabetes clinic-based survey. Diabetes Care. 2006 Dec;29(12):2701-7. doi: 10.2337/dc06-0942. PMID 17130208
- [Background] Lin SX, Pi-Sunyer EX. Prevalence of the metabolic syndrome among US middle-aged and older adults with and without diabetes--a preliminary analysis of the NHANES 1999-2002 data. Ethn Dis. 2007 Winter;17(1):35-9. PMID 17274207
- [Background] Yadav D, Mahajan S, Subramanian SK, Bisen PS, Chung CH, Prasad GB. Prevalence of metabolic syndrome in type 2 diabetes mellitus using NCEP-ATPIII, IDF and WHO definition and its agreement in Gwalior Chambal region of Central India. Glob J Health Sci. 2013 Sep 17;5(6):142-55. doi: 10.5539/gjhs.v5n6p142. PMID 24171882
- [Background] Song SH, Hardisty CA. Diagnosing metabolic syndrome in type 2 diabetes: does it matter? QJM. 2008 Jun;101(6):487-91. doi: 10.1093/qjmed/hcn034. Epub 2008 Mar 19. PMID 18353792
- [Background] Didangelos TP, Thanopoulou AK, Bousboulas SH, Sambanis CL, Athyros VG, Spanou EA, Dimitriou KC, Pappas SI, Karamanos BG, Karamitsos DT. The ORLIstat and CArdiovascular risk profile in patients with metabolic syndrome and type 2 DIAbetes (ORLICARDIA) Study. Curr Med Res Opin. 2004 Sep;20(9):1393-401. doi: 10.1185/030079904125004466. PMID 15383188
- [Background] Bo S, Ciccone G, Baldi C, Benini L, Dusio F, Forastiere G, Lucia C, Nuti C, Durazzo M, Cassader M, Gentile L, Pagano G. Effectiveness of a lifestyle intervention on metabolic syndrome. A randomized controlled trial. J Gen Intern Med. 2007 Dec;22(12):1695-703. doi: 10.1007/s11606-007-0399-6. Epub 2007 Oct 6. PMID 17922167
- [Background] Christensen P, Bliddal H, Riecke BF, Leeds AR, Astrup A, Christensen R. Comparison of a low-energy diet and a very low-energy diet in sedentary obese individuals: a pragmatic randomized controlled trial. Clin Obes. 2011 Feb;1(1):31-40. doi: 10.1111/j.1758-8111.2011.00006.x. PMID 25586973
- [Background] Yoon NH, Yoo S, Kim H, Han Y. Routine Screening and Consultation Facilitate Improvement of Metabolic Syndrome. J Korean Med Sci. 2015 Aug;30(8):1092-100. doi: 10.3346/jkms.2015.30.8.1092. Epub 2015 Jul 15. PMID 26240487
- [Background] Sharip, A., Firek, A., & Tonstad, S. The Effects of Smoking Cessation on the Risk Factors for the Metabolic Syndrome: A Follow-Up Study of Veterans. Journal of Smoking Cessation 2017, 12(3), 143-152. doi:10.1017/jsc.2016.10
- [Background] Polosa R, Morjaria JB, Caponnetto P, Battaglia E, Russo C, Ciampi C, Adams G, Bruno CM. Blood Pressure Control in Smokers with Arterial Hypertension Who Switched to Electronic Cigarettes. Int J Environ Res Public Health. 2016 Nov 11;13(11):1123. doi: 10.3390/ijerph13111123. PMID 27845734
- [Background] Polosa R, Morjaria JB, Caponnetto P, Caruso M, Campagna D, Amaradio MD, Ciampi G, Russo C, Fisichella A. Persisting long term benefits of smoking abstinence and reduction in asthmatic smokers who have switched to electronic cigarettes. Discov Med. 2016 Feb;21(114):99-108. PMID 27011045
- [Background] Polosa R, Morjaria JB, Prosperini U, Russo C, Pennisi A, Puleo R, Caruso M, Caponnetto P. Health effects in COPD smokers who switch to electronic cigarettes: a retrospective-prospective 3-year follow-up. Int J Chron Obstruct Pulmon Dis. 2018 Aug 22;13:2533-2542. doi: 10.2147/COPD.S161138. eCollection 2018. PMID 30197510
- [Background] Adriaens K, Van Gucht D, Declerck P, Baeyens F. Effectiveness of the electronic cigarette: An eight-week Flemish study with six-month follow-up on smoking reduction, craving and experienced benefits and complaints. Int J Environ Res Public Health. 2014 Oct 29;11(11):11220-48. doi: 10.3390/ijerph111111220. PMID 25358095
- [Background] Polosa R, Caponnetto P, Maglia M, Morjaria JB, Russo C. Success rates with nicotine personal vaporizers: a prospective 6-month pilot study of smokers not intending to quit. BMC Public Health. 2014 Nov 8;14:1159. doi: 10.1186/1471-2458-14-1159. PMID 25380748
- [Background] Pocock SJ. Clinical Trials: A practical approach. Wiley 1983
- [Background] Mann JFE, Orsted DD, Brown-Frandsen K, Marso SP, Poulter NR, Rasmussen S, Tornoe K, Zinman B, Buse JB; LEADER Steering Committee and Investigators. Liraglutide and Renal Outcomes in Type 2 Diabetes. N Engl J Med. 2017 Aug 31;377(9):839-848. doi: 10.1056/NEJMoa1616011. PMID 28854085
- [Background] Green JB, Bethel MA, Armstrong PW, Buse JB, Engel SS, Garg J, Josse R, Kaufman KD, Koglin J, Korn S, Lachin JM, McGuire DK, Pencina MJ, Standl E, Stein PP, Suryawanshi S, Van de Werf F, Peterson ED, Holman RR; TECOS Study Group. Effect of Sitagliptin on Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2015 Jul 16;373(3):232-42. doi: 10.1056/NEJMoa1501352. Epub 2015 Jun 8. PMID 26052984
- [Background] Marso SP, Bain SC, Consoli A, Eliaschewitz FG, Jodar E, Leiter LA, Lingvay I, Rosenstock J, Seufert J, Warren ML, Woo V, Hansen O, Holst AG, Pettersson J, Vilsboll T; SUSTAIN-6 Investigators. Semaglutide and Cardiovascular Outcomes in Patients with Type 2 Diabetes. N Engl J Med. 2016 Nov 10;375(19):1834-1844. doi: 10.1056/NEJMoa1607141. Epub 2016 Sep 15. PMID 27633186
- [Background] Buckley JP, Sim J, Eston RG, Hession R, Fox R. Reliability and validity of measures taken during the Chester step test to predict aerobic power and to prescribe aerobic exercise. Br J Sports Med. 2004 Apr;38(2):197-205. doi: 10.1136/bjsm.2003.005389. PMID 15039259
- [Background] Bradley C, Todd C, Gorton T, Symonds E, Martin A, Plowright R. The development of an individualized questionnaire measure of perceived impact of diabetes on quality of life: the ADDQoL. Qual Life Res. 1999;8(1-2):79-91. doi: 10.1023/a:1026485130100. PMID 10457741
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Florez H, Temprosa MG, Orchard TJ, Mather KJ, Marcovina SM, Barrett-Connor E, Horton E, Saudek C, Pi-Sunyer XF, Ratner RE, Goldberg RB; Diabetes Prevention Program Research Group. Metabolic syndrome components and their response to lifestyle and metformin interventions are associated with differences in diabetes risk in persons with impaired glucose tolerance. Diabetes Obes Metab. 2014 Apr;16(4):326-33. doi: 10.1111/dom.12220. Epub 2013 Oct 29. PMID 24118860
- [Derived] Krysinski A, Russo C, John S, Belsey JD, Campagna D, Caponnetto P, Vudu L, Lim CW, Purrello F, Di Mauro M, Iqbal F, Fluck D, Franek E, Polosa R, Sharma P; DIASMOKE collaborators. International randomised controlled trial evaluating metabolic syndrome in type 2 diabetic cigarette smokers following switching to combustion-free nicotine delivery systems: the DIASMOKE protocol. BMJ Open. 2021 Apr 27;11(4):e045396. doi: 10.1136/bmjopen-2020-045396. PMID 33906842
- See also: Standards of medical care in diabetes--2015: summary of revisions. Diabetes Care 38: S4, 2015 (pages 162-64) — http://aemmedi.it/wp-content/uploads/2018/06/AMD-Standard-unico-protetto.pdf
- See also: . McNeill A, Brose L S, Calder R, Bauld L and Robson D. Evidence review of e-cigarettes and heated tobacco products 2018. A report commissioned by Public Health England. — https://www.gov.uk/government/publications/e-cigarettes-and-heated-tobacco-products-evidence-review